CLINICAL TRIAL: NCT02287259
Title: A Randomized, Open Label Trial of Olanzapine Versus Lithium in the Treatment of Acute Depression in Patients With Bipolar II or Bipolar Not Otherwise Specified.
Brief Title: Olanzapine Versus Lithium in the Treatment of Acute Depression in Patients With Bipolar II or Bipolar Not Otherwise Specified(OL Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tadashi Hasegawa (Other)
Responsible Party: Sponsor-Investigator, Tadashi Hasegawa, medical doctor(assistant professor), Chiba University
Organization: Chiba University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChibaU
Record Dates: First submitted 2014-10-30; First posted 2014-11-10 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine; Lithium

ARMS (2):
- Olanzapine (Experimental): PO start with 2.5mg daily once for 7days, since then flexible dose.
  Interventions: Drug: olanzapine
- Lithium (Active Comparator): PO start with 400mg daily twice for 7days, since then flexible dose.
  Interventions: Drug: lithium

INTERVENTIONS:
Drug: olanzapine
  Arms: Olanzapine
Drug: lithium
  Arms: Lithium

SUMMARY:
Determine the efficacy and tolerability of olanzapine for treatment of acute depression in patients with bipolar II or bipolar disorder NOS compared with lithium.

ELIGIBILITY:
Inclusion Criteria:

* major depressive episode in type2 bipolar disorder or bipolar disorder NOS.(MADRS more than 20 point)
* 18years to 65years
* subjects who sign the informed consent document

Exclusion Criteria:

* don't have Diabetes and abnormal metabolism of sugar
* not noticed as bipolar disorder
* have an organic brain disease
* pregnant or breastfeeding women
* don't have heart disease
* have actively suicidal thought(Suicidal ideation score of MADRS is 6)
* who are judged by the investigator to should be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery- Åsberg Depression Rating(MADRS) | Baseline and 8 weeks

SECONDARY OUTCOMES:
Change in Young Mania Rating Scale(YMARS) | Baseline and 8 weeks
Quick Inventory of Depressive Symptomatology Japanese version(QIDS-J) | Baseline and 8 weeks
State Trait Anxiety Inventory Form JYZ(STAI) | Baseline and 8 weeks
Clinical Global Impression for Bipolar Disorder(CGI-BP) | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chiba University Hospital, Chiba, Japan